CLINICAL TRIAL: NCT01842256
Title: A Randomized, Open-label, Single Dose, Two-treatment, Two-period, Two-sequence Crossover Study to Investigate the Effect of Telmisartan/S-amlodipine on the Pharmacokinetic Properties of Atorvastatin After Oral Administration in Healthy Volunteers
Brief Title: Study to Investigate the Effect of Telmisartan/S-amlodipine on the Pharmacokinetic Properties of Atorvastatin.
Acronym: CKD-345
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 142HPS13002
Record Dates: First submitted 2013-04-25; First posted 2013-04-29 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Essential Hypertension; Hyperlipidemia
Keywords: Telminouveau; Atorvastatin; Pharmacokinetic; Healthy volunteers
MeSH Terms: conditions — Essential Hypertension; Hyperlipidemias | interventions — Telmisartan; levamlodipine; Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telmisartan 80mg, S-amlodipine 5mg and Atorvastatin 40mg (Experimental)
  Interventions: Drug: Telmisartan 80mg, S-amlodipine 5mg and Atorvastatin 40mg; Drug: atorvastatin 40mg
- Atorvastatin 40mg (Active Comparator)
  Interventions: Drug: Telmisartan 80mg, S-amlodipine 5mg and Atorvastatin 40mg; Drug: atorvastatin 40mg

INTERVENTIONS:
Drug: Telmisartan 80mg, S-amlodipine 5mg and Atorvastatin 40mg — * 3 Tablets (telmisartan 80mg, amlodipine 5mg, atorvastatin 40mg each one),
  * oral intake, once in a period
  * over the period Ⅰ&Ⅱ(crossover)
Drug: atorvastatin 40mg — * 1 Tablet (atorvastatin 40mg),
  * oral intake, once in a period
  * over the period Ⅰ&Ⅱ(crossover)

SUMMARY:
The purpose of this study is to investigate the effect of telmisartan/s-amlodipine on the pharmacokinetic properties of atorvastatin.

DETAILED DESCRIPTION:
healthy subjects are administrated single-dose over the period Ⅰand Ⅱ(Crossover) of telmisartan/s-amlodipine, atorvastatin and atorvastatin.

ELIGIBILITY:
Inclusion Criteria:

1. Between 20 aged and 45 aged in healthy male and female
2. Body weight more than 55kg in male, 50kg in female
3. Body Mass Index more than 18.5 and under 25 (Body Mass Index(kg/m2)= kg/(m)2)
4. If female, must include more than one among the items

   1. The menopause (there is no natural menses for at least 2 years)
   2. Surgical Infertility(hysterectomy or bilateral oophorectomy, tubal ligation or other methods of infertility condition)
   3. The male partner infertility before screening (Demonstrated azoospermia after vasectomy)and if this man is the only partner of the female subject.
   4. you are using one of the following contraceptive measure for 3 months before screening, and Necessarily you agree that used continuously contraceptive measure during the clinical trial and for 1 month after the final dosing investigational product.(But, should not use a device of contraception or oral contraceptive drug that containing a hormonal caused telmisartan, s-amlodipine, atorvastatin calcium drug interactions during the clinical trials)

      * Abstinence.
      * Physical interrupt method (such as a condom, contraceptive diaphoretic or cervical cap)
   5. In case of women of childbearing age, the serum β-hCG pregnancy test is negative, and urine β-hCG test is negative before taking the investigational product.
5. If men has sexual life with women of childbearing age, Necessarily he agrees that use condoms during clinical trials and do not sperm donation during clinical trials and until one month after the final dosage of investigational products
6. Those who fully understand about this clinical trial after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent.

Exclusion Criteria:

1. Have clinically significant disease that hepatobiliary system(severe hepatic impairment, etc), kidney(severe renal impairment, etc.), nervous system, immune system, respiratory system, endocrine system,hemato-oncology disease, cardiovascular system (heart failure, etc.).or mental illness, or a history of mental disease.
2. Have a gastrointestinal disease history that can affect drug absorption (Crohn, ulcers, etc.) or surgery (except simple appendectomy or hernia surgery)
3. Hypersensitivity reaction to drug or clinically significant hypersensitivity reaction in the history of Investigational drugs (telmisartan, s-amlodipine or atorvastatin calcium) or additives
4. An impossible one who participates in clinical trial including screening tests(medical history taking, BP, physical examination, 12-lead ECG, blood & urine laboratory test result) within 28 days before the beginning of study treatment.
5. Defined by the following laboratory parameters:

   * AST, ALT> 1.25*upper limit of normal range
   * Total bilirubin > 1.5* upper limit of normal range
   * CPK > 1.5* upper limit of normal range
   * eGFR(using by MDRD method) < 60 mL/min/1.73m2
6. Sitting SBP > 150 mmHg or < 90 mmHg, Sitting DBP> 100 mmHg or < 50 mmHg , after 5minuts break.
7. Drug abuse or have a history of drug abuse showed a positive for the Triage TOX drug on urine.
8. Pregnant or lactating women.
9. A heavy caffeine consumer(caffeine>5cups/day), alcohol consumer(alcohol>210g/week), or smoker(cigarette>10cigarettes /day)
10. Subject takes ethical drug or herbal medicine within 14days, OTC within 7days before the beginning of study treatment but investigator determine that the taking drug affect this study or could affect the safety of the subjects.
11. Subject who takes inhibitors and inducers of drug metabolizing enzyme(Barbiturates etc.) within 30 days.
12. Taking foods containing grapefruit within 7 days before the beginning of study treatment(ex. Drinking containing grapefruit of 1L per a day or more within 7 days before the beginning of study treatment)
13. Subject who treated with any investigational drugs within 60days before the beginning of study treatment (However, biologicals applies for 90 days, but can be based on a more extended period of time by considering the half-life.
14. Previously donate whole blood within 60 days or component blood within 30days.
15. An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
16. Positive for Hepatitis B, Hepatitis C, HIV

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-04; Primary Completion 2013-05 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
In the steady state atorvastatin 40mg AUClast | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  AUClast: Area under the plasma concentration time curve from zero time until the last measurable concentration.
In the steady state atorvastatin 40mg Cmax | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  Cmax: maximum plasma drug concentration

SECONDARY OUTCOMES:
In the steady state atorvastatin 40mg AUCinf | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  AUCinf: Area Under the Concentration time curve from time zero to infinity
In the steady state atorvastatin 40mg Tmax | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  Tmax: Time to Cmax
In the steady state atorvastatin 40mg t1/2 | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  t1/2: Observed terminal elimination half-life
Number of participants with adverse events | From 1day to 17days
  * Evaluated safety parameters included: physical examination, vital sign, laboratory test, ECG
  * Adverse event monitoring
In the steady state Orthohydroxy-atorvastatin AUClast | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  AUClast: Area under the plasma concentration time curve from zero time until the last measurable concentration.
In the steady state Orthohydroxy-atorvastatin Cmax | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  Cmax: maximum plasma drug concentration
In the steady state Orthohydroxy-atorvastatin AUCinf | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  AUCinf: Area Under the Concentration time curve from time zero to infinity
In the steady state Orthohydroxy-atorvastatin Tmax | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  Tmax: Time to Cmax
In the steady state Orthohydroxy-atorvastatin t1/2 | 0, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 36, 48hr post-dose
  t1/2: Observed terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Min Soo Park, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea